CLINICAL TRIAL: NCT06218108
Title: Multicenter Observational Study on the Taulí-T1 Classification for Staging, Prognosis, and Management of pT1 Rectal Adenocarcinoma (TAUTEM-pT1 Study)
Brief Title: Multicenter Observational Study Taulí-T1 Classification for the Management of pT1 Rectal Adenocarcinoma
Acronym: TAUTEM-pT1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Head Colorectal Research Group, Corporacion Parc Tauli
Other Study IDs: TAUTEM-pT1
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer Stage I
Keywords: T1 Rectal Adenocarcinoma; Early invasive rectal adenocarcinoma; TEM; Submucosal invasion; Prognosis of T1 rectal adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Histological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Taulí-T1 versus conventional classifications — All the slides of each case will be reviewed, selecting the one that contains the most invasive section, and this will be digitized to take measurements in micrometers with greater precision. To measure the degree of infiltration, the measurement of residual healthy submucosa (hrSB) will be used, which is the distance between the point of greatest infiltration and the muscularis propria. The total thickness of the submucosa in the tumor area will also be measured, taking as a reference the muscularis of the mucosa or, in its absence, the surface of the lesion, to calculate the percentage of infiltration of the submucosa. This percentage will be calculated as the inverse percentage of invasion with respect to the hrSB: (total thickness of the submucosa - hrSB / total thickness of the submucosa) x 100. The qualitative categories will be obtained: sm1 (< 33.3%), sm2 (33.3% - 66.6%) and sm3 (> 66.6%). Measurements will be also taken in micrometers for the conventional classifications.

SUMMARY:
BACKGROUND: Rectal cancer is the sixth most common neoplasm in Spain. In the early stages (pT1-N0), the treatment of choice is transanal endoscopic microsurgery. Treatment may be expanded to radical surgery if there are poor prognostic factors for the presence of metastatic lymph nodes and a risk of recurrence (up to 29%). The most determining histopathological factor is the degree of submucosal invasion. There are different classical classifications to assess this invasion, which pose difficulties in establishing objective and reproducible measurements. Casalots et al. propose a new classification (Taulí-T1) based on the measurement of residual healthy submucosa (hrSB), hypothesizing that a greater amount of healthy submucosa correlates with a better prognosis. Results show less healthy submucosa in the recurrence group, with a trend towards statistical significance (p=0.09).

OBJECTIVE: To compare the Taulí-T1 classification with conventional quantitative classifications (Kitajima, Ueno) and qualitative classifications (sm1, sm2, and sm3 by Kudo and Kikuchi).

METHODOLOGY: A multicenter observational retrospective cohort study comparing the Taulí-T1 classification with classical classifications in 317 patients with stage pT1 rectal adenocarcinoma, following the STROBE guidelines. The main variable is the measurement of tumor invasion in µm through hrSB, compared to the invasion of quantitative (Kitajima and Ueno) and qualitative (Kudo and Kikuchi) classical classifications. Concordance will be assessed with the intraclass correlation coefficient for quantitative variables and Cohen's weighted kappa for qualitative variables, with a 95% confidence interval and p<0.005.

DETAILED DESCRIPTION:
HYPOTHESIS: Taulí-T1 classification will have greater clinical utility to classify the stage pT1 rectal adenocarcinomas compared with conventional classifications.

OBJECTIVE: The main objective of the study is to compare the Taulí-T1 classification versus the conventional quantitative methods (Kitajima, Ueno) and qualitative ones (sm1, sm2 and sm3 of Kudo and Kikuchi), through a multicenter cohort study of the TAUTEM group.

STUDY DESIGN:

Multicenter observational retrospective cohort study that compares the Taulí-T1 classification with the classic classifications for stage pT1 of rectal adenocarcinoma.

The study participants will be patients diagnosed with rectal cancer who underwent surgery using transanal endoscopic surgery technique (TME, TEO or TAMIS) and histopathologically diagnosed with stage pT1 rectal adenocarcinoma. To calculate the sample size, an alpha error of 0.05 was used with a confidence level of 95%, with a precision of 0.05 and an estimate of the prevalence of pT1 recurrence of 29%. A sample of 317 patients will be required.

The main variable to be studied is the measurement of tumor invasion in µm by measuring the healthy residual submucosa (hrSB) with the Taulí-T1 classification, in comparison with the measurement of invasion of the classic quantitative (Kitajima and Ueno) and qualitative classifications (Kudo and Kikuchi).

The secondary variables to be assessed are: demographic and macroscopic data of the tumor and histopathological variables (tumor morphology, measurement of the submucosa in the area of the lesion and in the healthy area, presence or absence of muscularis mucosa and muscularis propria, assessment of resection margins, histological differentiation degree, presence of adenocarcinoma on adenoma, presence of poor prognostic factors -lymphatic, perineural and vascular invasion, tumor budding-). Surgical data will also be collected (type of surgery, location of the tumor and distance from the anal margin, integrity of the specimen) and clinical data (neoadjuvant treatment, recurrences, appearance of lymphadenopathy, survival).

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma.
* Histopathologically diagnosed with stage pT1.
* Patients treated with transanal endoscopic surgery technique (TME, TEO or TAMIS).
* Patients who have received prior neoadjuvant treatment (radiotherapy and/or chemotherapy).
* Over 18 years.

Exclusion Criteria:

* Patients treated with other surgical techniques other than transanal endoscopic surgery.
* Tumors other than adenocarcinoma.
* Locations other than rectum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients diagnosed with rectal cancer who underwent surgery using transanal endoscopic surgery technique (TME, TEO or TAMIS) and histopathologically diagnosed with stage pT1 rectal adenocarcinoma. Patients who have received prior neoadjuvant treatment (radiotherapy and/or chemotherapy) will also be included, but both histological findings and their recurrence and survival data will be analyzed separately.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Taulí-T1 versus conventional classifications | 30 days
  Compare the Taulí-T1 classification versus the conventional quantitative methods (Kitajima, Ueno) and qualitative ones (sm1, sm2 and sm3 of Kudo and Kikuchi), to classify the stage pT1 rectal adenocarcinomas.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Hospital Universitario Parc Tauli de Sabadell, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casalots A, Serra-Aracil X, Mora-Lopez L, Garcia-Nalda A, Pericay C, Ferreres JC, Navarro-Soto S. T1 Rectal Adenocarcinoma: a Different Way to Measure Tumoral Invasion Based on the Healthy Residual Submucosa with Its Prognosis and Therapeutic Implications. J Gastrointest Surg. 2021 Oct;25(10):2660-2667. doi: 10.1007/s11605-021-04948-9. Epub 2021 Feb 24. PMID 33629231
- [Derived] Gener-Jorge C, Ferreres Pinas JC, Moreno Garcia AB, Melgar Rivera DS, Casalots A, Nonell A, Espina B, Caro-Tarrago A, Serra-Aracil X. Interobserver agreement of the Tauli-pT1 classification in rectal pT1 adenocarcinoma. Int J Colorectal Dis. 2025 Sep 17;40(1):201. doi: 10.1007/s00384-025-04996-6. PMID 40957973